CLINICAL TRIAL: NCT07151352
Title: Footwear and Brain Activity in Children: Insights From EEG During Walking
Brief Title: Footwear and Brain Activity in Children
Acronym: FooTBAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Gabriel Gijon-Nogueron, Professor, University of Malaga
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UCCSSMalaga
Record Dates: First submitted 2025-08-15; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Foot; Footwear; Children
Keywords: Children; footwear; Gait; electroencephalography

STUDY DESIGN:
Intervention Model Description: This is a within-subject, randomized crossover study in which each participant will complete a walking task under three different footwear conditions: barefoot, barefoot-style (minimalist) shoes, and conventional shoes with heel drop. The order of the conditions will be randomized for each participant to minimize order effects and fatigue. All participants will serve as their own controls, allowing direct comparison of cortical activity across conditions. Each walking trial will be performed on the same 10-meter walkway, with rest periods between conditions to reduce carryover effects.
Who Masked: Outcomes Assessor
Masking Description: This study will be conducted as an open-label trial with no masking. Due to the visible nature of the footwear conditions (barefoot, barefoot-style, and conventional shoes with heel drop), neither participants nor investigators can be blinded to the assigned condition during each walking trial. Data analysts will receive de-identified EEG datasets labeled only by condition codes to minimize potential bias during statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Starting Condition - Barefoot (Sham Comparator): Participants will first complete the walking task barefoot along a 10-meter walkway. They will then perform the same task in barefoot-style (minimalist) footwear and in conventional footwear with heel drop. The order of the second and third conditions will be randomized. EEG will be recorded during all walking trials, with rest periods between conditions.
  Interventions: Other: Starting Condition - Barefoot; Other: Barefoot-Style Footwear; Other: Conventional Footwear with Heel Drop
- Starting Condition - Barefoot-Style Footwear (Experimental): Participants will first complete the walking task in barefoot-style (minimalist) footwear with a 3 mm flexible sole, 0 mm heel drop, wide toe box, and no rigid heel counter. They will then perform the task barefoot and in conventional footwear with heel drop. The order of the second and third conditions will be randomized. EEG will be recorded during all walking trials, with rest periods between conditions.
  Interventions: Other: Starting Condition - Barefoot; Other: Barefoot-Style Footwear; Other: Conventional Footwear with Heel Drop
- Starting Condition - Conventional Drop Footwear (Active Comparator): Participants will first complete the walking task in conventional structured footwear with a rigid sole (12 mm heel / 7 mm forefoot), 5 mm heel drop, reinforced heel counter, and narrow toe box. They will then perform the task barefoot and in barefoot-style footwear. The order of the second and third conditions will be randomized. EEG will be recorded during all walking trials, with rest periods between conditions.
  Interventions: Other: Starting Condition - Barefoot; Other: Barefoot-Style Footwear; Other: Conventional Footwear with Heel Drop

INTERVENTIONS:
Other: Starting Condition - Barefoot — Participants walk barefoot along a 10-meter walkway without wearing shoes or socks.
  Other Names: No Shoes
Other: Barefoot-Style Footwear — Participants walk along a 10-meter walkway wearing minimalist footwear with a 3 mm flexible sole, 0 mm heel drop, wide toe box, and no rigid heel counter.
  Other Names: Minimalist shoes
Other: Conventional Footwear with Heel Drop — Participants walk along a 10-meter walkway wearing structured footwear with a rigid sole (12 mm heel / 7 mm forefoot), 5 mm heel drop, reinforced heel counter, and narrow toe box.
  Other Names: Structured shoes

SUMMARY:
Childhood is a critical period for neuromotor development, during which footwear may influence both gait biomechanics and the integration of sensory and motor control processes. This study will aim to analyze brain activity in children aged 6-7 years while walking under three conditions: barefoot, in barefoot-style (minimalist) shoes, and in conventional shoes with heel drop.

A quasi-experimental, repeated-measures study will be conducted, in which each participant will complete a 10-meter walking task under the three conditions, in randomized order. Brain activity will be recorded using a 14-channel wireless electroencephalography (EEG) system (Emotiv EPOC X), and relative spectral power (theta, alpha, beta, gamma) as well as Theta/Alpha and Beta/Alpha ratios will be calculated.

Statistical analysis will include global and regional comparisons (frontal, temporal, parieto-occipital), assessment of hemispheric asymmetry, and multivariate analysis. The study is expected to provide novel information on how footwear type may modulate cortical organization during children's gait, with potential implications for pediatric footwear design and clinical recommendations.

DETAILED DESCRIPTION:
Background and Rationale Between the ages of 5 and 8 years, basic movement patterns are consolidated and brain plasticity reaches one of its highest levels. Footwear, as an external factor, may modify both gait mechanics and the quality of sensory input reaching the central nervous system. Previous studies suggest that barefoot walking or minimalist footwear may enhance intrinsic foot muscle activation and proprioception; however, limited evidence exists on how these conditions affect cortical activity in children. Electroencephalography (EEG) offers a non-invasive and real-time method to record brain activity during motor tasks, making it a suitable tool for investigating this phenomenon.

Primary Objective The primary objective will be to analyze cortical activity using EEG in children aged 6-7 years while walking under three conditions: barefoot, in barefoot-style footwear, and in conventional footwear with heel drop.

Study Design A quasi-experimental, repeated-measures, within-subject design will be used. Each participant will be assessed under all three experimental conditions, with the order randomized to minimize learning or fatigue effects.

Participants The study will include 37 healthy children aged 6 to 7 years, with no neurological or musculoskeletal disorders, normal motor development, and no habitual use of barefoot-style footwear in the past six months.

Procedure

Each participant will walk 10 meters in three conditions:

Barefoot

Barefoot-style footwear (3 mm sole, flexible, 0 mm drop, wide toe box)

Conventional footwear with heel drop (rigid sole, 12 mm heel / 7 mm forefoot, 5 mm drop, reinforced heel counter, narrow toe box).

Brain activity will be recorded using the Emotiv EPOC X wireless EEG system (14 channels) and analyzed using EEGLAB (MATLAB). Relative power in theta (4-7 Hz), alpha (8-12 Hz), beta (13-30 Hz), and gamma (30-45 Hz) frequency bands will be calculated, along with Theta/Alpha and Beta/Alpha ratios.

Statistical Analysis A repeated-measures ANOVA and Tukey's post-hoc tests will be applied to compare conditions. Regional analysis, hemispheric asymmetry evaluation, and multivariate analyses (PCA, LDA) will also be performed. Statistical significance will be set at p < 0.05.

Expected Impact This study is expected to improve understanding of how footwear type influences cortical organization during children's gait. Findings may help inform pediatric footwear design and clinical recommendations to support healthy neuromotor development.

Ethics and Consent The protocol has been approved by the Ethics Committee of the University of Málaga (CEUMA112104). Written informed consent will be obtained from parents or legal guardians, and verbal assent will be obtained from all child participants.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-7 years.
* Typical motor and neurological development according to school or medical reports.
* Ability to understand and follow simple instructions.
* No regular use of barefoot-style footwear in the past six months.
* Written informed consent provided by a parent or legal guardian.
* Verbal assent provided by the child in an age-appropriate manner.

Exclusion Criteria:

* Diagnosed neurodevelopmental disorders (e.g., ADHD, autism spectrum disorder, motor dysfunction).
* Orthopedic or neuromuscular conditions affecting gait (e.g., equinus foot, cerebral palsy).
* Lower-limb surgery within the previous 6 months.
* Use of medication affecting alertness, muscle tone, or motor control.
* Scalp lesions or intolerance to EEG headset use.
* Any condition that, in the investigator's judgment, could interfere with study participation or data integrity.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Relative spectral power ratios (Theta/Alpha, Beta/Alpha) during walking in children | Day 1 (single data collection session)
  EEG-based measurement of relative spectral power in theta (4-7 Hz), alpha (8-12 Hz), and beta (13-30 Hz) frequency bands, and calculation of Theta/Alpha and Beta/Alpha ratios across three footwear conditions (barefoot, barefoot-style, conventional with heel drop). EEG will be recorded using a 14-channel Emotiv EPOC X system during a 10-meter walking task. Analyses will compare regional and global cortical activity patterns between conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaga, Málaga, Malaga, Spain

IPD SHARING:
Plan to Share IPD: No